CLINICAL TRIAL: NCT00692458
Title: A Phase III Study to Assess the Safety, Tolerability, and Efficacy of MK0822 (Odanacatib) in Reducing the Risk of Bone Metastasis in Women With Breast Cancer
Brief Title: A Study to Assess the Effects of MK0822 in Reducing the Risk of Bone Metastasis in Women With Breast Cancer (0822-029)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn for administrative reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0822-029; 2008_526; MK-0822-029
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): odanacatib
  Interventions: Drug: Comparator: odanacatib
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: Comparator: odanacatib — odanacatib; 5mg oral, once daily for approximately 60 months.
  Arms: 1
Drug: Comparator: placebo — placebo; oral, once daily for approximately 60 months
  Arms: 2

SUMMARY:
The purpose of this study is to test MK0822 on reducing the risk of bone metastasis in women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary State II or Stage III breast cancer
* Patient is not receiving adjuvant chemotherapy (e.g., cyclophosphamide, doxorubicin, carboplatin) at the time of randomization and has not received adjuvant chemotherapy for at least 6 weeks prior to the randomization visit (Visit 2). This inclusion criterion does not include hormone therapy, which is permitted (see inclusion criterion # 7)
* Patient is not receiving hormonal therapy OR if patient is receiving hormonal therapy (e.g., leuprolide, tamoxifen, anastrozole) she is on a stable regimen for at least 3 months at the time of screening (Visit 1). If patient is HER2-positive and is receiving trastuzumab treatment, she must be on a stable regimen for at least 1 month at the time of Visit 1
* Patient is not pregnant or breast-feeding. All women of childbearing potential must have a negative urine pregnancy test at screening (Visit 1)

Exclusion Criteria:

* Bone metastases or history of bone metastases
* Patient has evidence of other distant metastases (e.g., visceral, soft-tissue, or brain)
* Patient has had a prior local or regional recurrence of her breast cancer, or a contralateral tumor. DCIS (ductal carcinoma in-situ), and LCIS (local carcinoma in-situ) in either the ipsilateral or contralateral breast are permitted
* Patient has ANY of the following:

  1. is currently receiving a bisphosphonate or other drug therapy for osteoporosis
  2. has been treated with an oral bisphosphonate for osteoporosis for more than 3 months within the 2 years prior to Visit 1, or for a total of more than 6 months at any time prior to Visit 1
  3. has been treated with an intravenous bisphosphonate within the 12 months prior to Visit 1
* Patient has a history of malignancy other than breast cancer <5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Patients with melanoma, leukemia, lymphoma, and myeloproliferative disorders of any duration are exclusionary
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of signing the informed consent
* Patient is currently participating in or has at any time in the past participated in a breast cancer study with a registered medication (i.e., approved by the regulatory agency in which she resides) being tested for the treatment of breast cancer (an unapproved indication)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
to assess the effect of treatment with MK0822 5 mg once daily on the risk of developing a first bone metastasis compared to placebo | approximately 60 months (event driven study)

SECONDARY OUTCOMES:
to assess the effect of treatment with MK0822 5 mg once daily on disease-free survival compared to placebo | approximately 60 months (event driven study)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC